CLINICAL TRIAL: NCT02618655
Title: Clinical Research for the Diagnosis of Tick-borne Diseases in Patients With Unexplained Acute Fever
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Collaborators: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Fu Xueying, Clinical Research for the Diagnosis of Tick-borne Diseases in Patients With Unexplained Acute Fever, Beijing Friendship Hospital
Other Study IDs: Z151100004015029
Record Dates: First submitted 2015-11-28; First posted 2015-12-01 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Fever of Unknown Origin; Tick-borne Diseases
Keywords: TBDs；diagnosis
MeSH Terms: conditions — Fever of Unknown Origin; Tick-Borne Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Biospecimen Retention: Samples With DNA — whole blood, serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Fever，none definite diagnosis: Those who have fever，but the doctor can not make definite diagnoses with the diagnostic methods available.
  Interventions: Other: diagnostic methods

INTERVENTIONS:
Other: diagnostic methods — explore several laboratory diagnostic methods to find out which will be more helpful for making an accurate diagnosis in the early period of TBDs.

SUMMARY:
The study will use several laboratory diagnoses in the diagnosis of patients with fever，to find out which will be more helpful for making an accurate diagnosis in the early period of Tickborne Diseases.

DETAILED DESCRIPTION:
Tickborne Diseases(TBDs) spread throughout many countries and regions. In recent years, the incidence has a tendency to rise continuously. The clinical symptoms and laboratory features of tick-borne diseases are always of no specific, and the diagnostic methods available, such as observing the pathogen after cultivation or by the method of Gimenez、serological tests for antibody always can't make a timely diagnosis, especially in the early period of the disease. The development of polymerase chain reaction(PCR) has been applied for pathogen detection, and showed high sensitivity and specificity,and may contribute to early diagnose，but no standardized method of PCR has been as yet proposed. This study mean to explore several laboratory diagnoses to find out which will be more helpful for making an accurate diagnosis in the early period of TBDs.

ELIGIBILITY:
Inclusion Criteria:

* patients have fever more than one week
* temperature is higher than 38℃ Celsius degree
* full of physical examination and laboratory examination have been carried out after one week，but still cannot make a definite diagnosis

Exclusion Criteria:

* fever for non-infectious diseases such as rheumatic autoimmune disease or with tumor
* we find that the patient selected does not meet the selection criteria within the observation period
* patients leave with automatic discharge

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all the people who have fever with unknown origin
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-03; Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Evidence of immunoglobulin M and immunoglobulin G titres in acute and convalescent serum or a fragment of the specific gene from patients' whole blood | within the first 14 days in hospital

SECONDARY OUTCOMES:
the sensitivity and specificity of the laboratory diagnostic methods Related to the reserach | up to three years
  compare the sensitivity and specificity of all the laboratory diagnostic methods, using statistical methods, to find out the most helpful one for making an accurate diagnosis in the early period of TBDs.

CONTACTS AND LOCATIONS:
Overall Officials: wenjie Qi, archiater, Study Director — Beijing Friendship Hospital
Locations (1):
- Organization Name Beijing Friendship Hospital,Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes